CLINICAL TRIAL: NCT06997601
Title: Serratus Posterior Superior Intercostal Plane Block Versus Suprascapular Nerve Block and Axillary Nerve Block for Analgesia in Shoulder Arthroscopic Surgery: A Randomized Clinical Trial
Brief Title: Serratus Posterior Superior Intercostal Plane Block Versus Suprascapular Nerve Block and Axillary Nerve Block for Analgesia in Shoulder Arthroscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSharkawy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264PR1191/4/25
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Serratus Posterior Superior Intercostal Plane Block; Suprascapular Nerve Block; Axillary Nerve Block; Analgesia; Shoulder Arthroscopic Surgery
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group SPSIPB (Experimental): Patients will receive a serratus posterior superior intercostal plane block.
  Interventions: Other: Serratus posterior superior intercostal plane block
- Group SSSB+ANB (Experimental): Patients will receive suprascapular nerve block + axillary nerve block.
  Interventions: Other: Suprascapular nerve block + Axillary nerve block

INTERVENTIONS:
Other: Serratus posterior superior intercostal plane block — Patients will receive a serratus posterior superior intercostal plane block.
  Arms: Group SPSIPB
Other: Suprascapular nerve block + Axillary nerve block — Patients will receive suprascapular nerve block + axillary nerve block.
  Arms: Group SSSB+ANB

SUMMARY:
This study aims to compare the serratus posterior superior intercostal plane block and suprascapular nerve block and axillary nerve block for analgesia in shoulder arthroscopic surgery.

DETAILED DESCRIPTION:
Controlling postoperative pain while minimizing opioid administration is particularly important because poor pain control is thought to be responsible for more than 60% of unplanned or prolonged hospitalizations.

Suprascapular nerve block (SSNB) has been proposed based on the anatomic fact that the suprascapular nerve innervates approximately 70% of the shoulder joint, capsule, subacromial space, acromioclavicular joint, and coracoacromial ligament, with the remaining 30% thought to be innervated by the lateral pectoral and axillary nerve.

The combined SSNB and axillary nerve block (ANB) was proposed as a safe alternative to interscalene brachial plexus block (ISB) for providing anesthesia and postoperative analgesia for shoulder surgery.

Serratus posterior superior intercostal plane block (SPSIPB) was described as a novel technique in a case series study of cadavers and five patients.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years.
* Both sexes.
* American Society of Anesthesiology (ASA) physical status I-II.
* Scheduled for open thoracotomy.

Exclusion Criteria:

* Infection at the site of regional blocks.
* Allergy to any drug used in this study.
* Use of psychotropic and/or narcotic medications on a regular basis.
* Cognitive dysfunction.
* Cardiovascular disease.
* Pulmonary disease.
* Coagulation abnormalities.
* Anatomical abnormalities.
* Neuropathic pain.
* Body mass index >40.
* History of substance abuse.
* Previous surgery in the same shoulder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2025-05-31 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Time to the 1st rescue analgesia | 24 hours postoperatively
  Time to the first request for the rescue analgesia (time from end of surgery to first dose of morphine administered).

SECONDARY OUTCOMES:
Degree of pain | 24 hours postoperatively
  Each patient will be instructed about postoperative pain assessment with the numeric rating scale (NRS) score. NRS (0 represents "no pain" while 10 represents "the worst pain imaginable"). NRS will be assessed at 0, 2, 4, 6, 8, 12, 18, and 24 h postoperatively.
Intraoperative fentanyl consumption | Intraoperatively
  Additional fentanyl bolus dosages of 1 µg/kg IV will be administered if the heart rate or mean arterial blood pressure is elevated by more than 20% of the baseline.
Total morphine consumption | 24 hours postoperatively
  Rescue analgesia of morphine will be given as 3 mg bolus if the numeric rating scale (NRS)> 3 to be repeated after 30 min if pain persists until the NRS < 4.
Incidence of adverse events | 24 hours postoperatively
  Incidence of adverse events such as bradycardia, hypotension, nausea, vomiting, respiratory depression, or any other complication.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.